CLINICAL TRIAL: NCT06550934
Title: Surgical Treatment of Pelvis in Fragility Fracture in Germany: a Prospective, National, Multicenter, Observational, Comparative Cohort Study Comparing Isolated Posterior Versus Combined Anterior-posterior Surgical Fracture Stabilization
Acronym: AO TOP
Status: Not yet recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Collaborators: AUC - Akademie der Unfallchirurgie (Unknown); AO Trauma Deutschland e.V. (Other)
Responsible Party: Sponsor
Other Study IDs: AO TOP
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pelvis; Fracture
Keywords: Pelvis; Fragility fracture; Classification; Management; Operative; Outcome
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Isolated posterior surgical fracture stabilization
  Interventions: Procedure: Fracture stabilization
- Combined anterior-posterior surgical fracture stabilization
  Interventions: Procedure: Fracture stabilization

INTERVENTIONS:
Procedure: Fracture stabilization — isolated posterior surgical fracture stabilization vs. combined anterior-posterior surgical fracture stabilization

SUMMARY:
Over a period of approximately two years, patients above the age of 65 who have suffered from an FFP equal to or higher than type IIc FFP, according to Rommens and Hofmann, will be eligible for inclusion. At least 420 patients will be included and followed up up for 12 months. Treatment and postoperative care, will be as per standard of care at the participating institution, with a free choice of isolated posterior or combined anterior-posterior surgical treatment.

Pain levels, quality of life, level of mobility and independence will be assessed at different time points. Furthermore, both clinical and radiographic outcomes, complications, morbidity and mortality associated with interventions will be evaluated. Assessment and evaluation will be performed at defined time points during FU according to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sacral FFP (no concomitant injuries) Types: IIc, IIIc, IVb, IVc according to Rommens and Hofmann associated with fracture of the anterior pelvic ring (fractures involving the anterior lip of the acetabulum that are not regarded as acetabular fracture will be included)
* Diagnostic workup for fracture diagnosis and classification performed using CT scan as per standard of care
* Indication for surgical fracture fixation as considered by the attending surgeon
* Age ≥ 65 yrs.
* Low-energy trauma fracture, or osteoporotic fracture, or insufficiency fracture, or spontaneous fracture
* ASA-Score ≤ 3 pts.
* Ability to provide informed consent according to the IRB/EC defined and approved procedures

Exclusion Criteria:

* Patients with multiple fractures
* Instability of the pubic symphysis (ie, visibility of a widening or diastasis of the symphysis), and/or fractures of the pubic rami next to the symphysis, that indicate instability
* Pelvic fractures due to high-energy trauma
* Pathologic fractures (eg, fractures caused by malignancy or infection)
* History of pelvic fracture or pelvic ring surgery (hip joint implants do not count)
* Clinically significant or unstable medical or surgical condition that prevents surgical treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 65 years or older with a fragility fracture in the pelvis.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Pain rating | Numeric Rating Scale (NRS) 3 month after surgical fixation of the fragility fracture of the pelvis
  Perception of pain will be assessed using Numeric Rating Scale (NRS) from 1-10, where patient reports pain due to his/her pelvis fracture. A higher value correlates with greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stange, Prof, Principal Investigator — Universitätsklinikum Münster; Lars Grossterlinden, Prof, Principal Investigator — Asklepios Klinik Altona, Hamburg

IPD SHARING:
Plan to Share IPD: No